CLINICAL TRIAL: NCT00886951
Title: Evaluation of [123I] MNI-388 and 123-I MNI-390 and SPECT as Markers of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Single Photon Emission Computed Tomography (SPECT) Imaging Study to Develop a Biomarker for Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: There seemed to be no uptake of the ligand in the areas of the brain expected for subjects with amyloid.
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-388/390-01
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access I123MNI388/I123MNI390 and brain imaging (Experimental)
  Interventions: Drug: I123MNI388/I123MNI390

INTERVENTIONS:
Drug: I123MNI388/I123MNI390 — Subjects will be dosed by intravenous injection up to 5 mCi and not to exceed 5.5 (not >10% of 5 mCi limit) 123-I MNI-388 or 123-I MNI-390.

SUMMARY:
The main objectives of this proposal are as follows:

* To assess the dynamic uptake and washout of 123-I MNI-388 and MNI 390, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in similarly aged Alzheimer's (AD) subjects and healthy controls
* To perform blood metabolite characterization of 123-I MNI-388 and MNI-390 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of 123-I MNI-388 and MNI 390 as a single photon computed tomography (SPECT) brain imaging agent

DETAILED DESCRIPTION:
The adaptation of imaging agents like 123-I MNI-388 and 123-I MNI-390 as biomarkers of β-amyloid deposition in AD patients for assessing disease requires human validation studies. The purpose of this study is to develop and characterize 123-I MNI-388 and 123-I MNI-390 as objective biomarkers in AD. The significance of this work lies in applying state-of-art quantitative neuroimaging tools to develop a relevant biomarker in living AD patients. In this context we propose to investigate the feasibility of applying this technique as an imaging biomarker of disease in AD patients.

Informed consent will be obtained for all subjects. All subjects will undergo a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be given a bolus injection of 123-I MNI-388 and MNI 390 in an antecubital vein. Subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I MNI-388 and MNI 390 in plasma (both protein bound and free) over a period of up to 8 hours. The quantitative and visual imaging analyses will be performed by an image-processing specialist who will remain blinded to any clinical information.including diagnosis. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-388 and MNI-390. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the AD patients and controls will be compared.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's Subject Selection: subjects who have a clinical diagnosis of mild to moderate Alzheimer's disease will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* CDR score ≥0.5 and <2.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-388 or 123-I MNI-390 injection.

Exclusion Criteria:

Alzheimer's subjects will be excluded from participation for the following reasons:

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Clinically significant MRI evidence of vascular disease or alternative neurologic disorder
* Pregnancy

Concomitant therapy: patients may remain on a stable dose of anticholinesterase medication during the study. Use of donepezil (Aricept®), rivastigmine (Exelon®), galantamine (Razadyne®), tacrine (Cognex®), and memantine (Namenda®) are permitted during the study. Doses of these compounds must be stable for 2 months prior to the study. At each visit after the screening visit, the investigator will ask the patient whether any medications including OTC medications, were taken since the previous visit.

Use of antipsychotics for agitation and benzodiazepines for insomnia or anxiety is permitted. However, the use of these agents is not permitted within the 8 hours prior to administration of cognitive testing.

Inclusion Criteria:

Healthy Control Subject Selection: Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* CDR score 0.
* For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-388 or 123-I MNI-390 injection.

Exclusion Criteria:

Healthy control subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has participated in another clinical study within the previous 30 days.
* Pregnancy
* Clinically significant MRI evidence of vascular disease or neurologic disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the reliability of MNI 388/390 as a potential imaging biomarker for amyloid imaging in the brain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States